CLINICAL TRIAL: NCT04009408
Title: Interventional Study of Expiratory Muscle Strength Training as a Treatment in Neuromuscular Disorders
Brief Title: Expiratory Muscle Strength Training (EMST) in Neuromuscular Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Calgary (Other)
Collaborators: Muscular Dystrophy Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REB18-1121
Record Dates: First submitted 2019-06-06; First posted 2019-07-05 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Oculopharyngeal Muscular Dystrophy; Muscular Dystrophies; Myopathy; Hereditary
Keywords: Dysphagia; Myopathy; Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Oculopharyngeal; Muscular Dystrophies; Muscular Diseases; Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: Parallel group, double blind, sham controlled study
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will not be informed until the end of study whether they received active intervention or sham intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- EMST therapy (Experimental): Participants use the EMST device as per study protocol, set to 50% of the patient's maximal expiratory pressure, as measured by handheld manometer.
  Interventions: Device: Expiratory muscle strength therapy (EMST150, Aspire LLC)
- Sham EMST therapy (Sham Comparator): Participants use a sham EMST device that has the spring removed as per study protocol, with no significant airflow resistance.
  Interventions: Device: Expiratory muscle strength therapy (EMST150, Aspire LLC)

INTERVENTIONS:
Device: Expiratory muscle strength therapy (EMST150, Aspire LLC) — Active therapy calibrated to the participant's maximum expiratory pressure

SUMMARY:
The purpose of this study is to investigate the impact of expiratory muscle strength training (EMST) on the swallowing, breathing, oral intake, quality of life and cough function of people with oculopharyngeal muscular dystrophy (OPMD).

DETAILED DESCRIPTION:
Outline:

Twenty participants with OPMD, with dysphagia, will be recruited from Neuromuscular clinics within Calgary. The investigators will enrol patients in a parallel group, sham-controlled, randomized clinical trial, with 10 participants in each group (active EMST and sham EMST).

Participants will have baseline measurements of: (i) global swallowing function via modified barium swallow study, (ii) maximum expiratory pressure, (iii) voluntary cough spirometry, (iv) forced vital capacity, (v) functional oral intake, (vi) patient report of self-perceived swallowing impairment (EAT-10 Questionnaire), and (vii) biomarker analyses.

Participants will undergo 5-weeks of EMST (active or sham). All baseline measurements will be repeated after 5-weeks of EMST and 10-weeks post-EMST to measure durability of effect.

Outcomes:

The end-goal of the current research is to obtain preliminary data for the benefit of EMST in a new study population, and direct future studies that may provide evidence for a new standard of care in treating neuromuscular diagnoses.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of oculopharyngeal muscular dystrophy (OPMD)
* 18 years of age or older
* Must be capable of providing informed consent
* Must be able to undergo respiratory function testing and swallowing studies
* Must have a forced vital capacity (FVC) greater than 60%
* A score of 3 or greater on the Eating Assessment Tool-10 (EAT-10; self-administered, symptom-specific outcome instrument for dysphagia. A score of 3 or greater indicates increased stress around eating)
* A score of 26 or greater on the Montreal Cognitive Assessment (MoCA; 30-point screening assessment used for detecting cognitive impairment. A score of 26 or greater is considered to be within functional limits.)

Exclusion Criteria:

* Severe coronary artery disease
* Acute myocardial infarction
* Moderate to severe hypovolemia
* Acute neurological events
* Unstable cardiac status
* Recent hernia
* Severe chronic obstructive pulmonary disease (COPD)
* Uncontrolled reflux issues
* Women who are pregnant, or who suspect they may be pregnant
* Cognitive impairment that would prevent comprehension of instructions and adherence to intervention guidelines (a score of less than 26 points on the MoCA)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Global Swallowing Function | Change in score from week 0 to week 5
  Global swallowing function is rated from videofluoroscopy swallowing studies (VFSS), using the Dynamic Imaging Grade of Swallowing Toxicity (DIGEST), a validated 5-point scale. Global swallowing function is rated from 0-4: 0 = no pharyngeal dysphagia; 1 = mild; 2 = moderate; 3 = severe; 4 = life-threatening. A lower score is a better outcome.

SECONDARY OUTCOMES:
Global Swallowing Function | Change in score from week 0 to week 15; change in score from week 5 to week 15.
  Global swallowing function is rated from videofluoroscopy swallowing studies (VFSS), using the Dynamic Imaging Grade of Swallowing Toxicity (DIGEST), a validated 5-point scale. Global swallowing function is rated from 0-4: 0 = no pharyngeal dysphagia; 1 = mild; 2 = moderate; 3 = severe; 4 = life-threatening.
Maximum expiratory pressure (MEP) | Change in score from week 0 to week 5; change in score from week 0 to week 15; change in score from week 5 to week 15.
  MEP is a measure of respiratory muscle strength and is assessed with a handheld manometer, measured in centimetres of water (cmH2O). A higher score is a better outcome.
Volitional cough strength (peak cough flow) | Change in score from week 0 to week 5; change in score from week 0 to week 15; change in score from week 5 to week 15.
  Measure of cough strength that is assessed using a spirometer, measured in litres per minute (L/min). A higher score is a better outcome.
Forced vital capacity (FVC) | Change in score from week 0 to week 5; change in score from week 0 to week 15; change in score from week 5 to week 15.
  Measure of how much air is exhaled during forced exhalation and is assessed with a spirometer, measured in litres. A higher score is a better outcome.
Oral Intake | Change in score from week 0 to week 5; change in score from week 0 to week 15; change in score from week 5 to week 15.
  A measure daily nutritional and hydration consumption. Oral intake is assessed using the Functional Oral Intake Scale (FOIS), a validated 7-point ordinal scale (1 = no oral intake; 2 = tube dependent with minimal/inconsistent oral intake; 3 = tube supplements with consistent oral intake; 4 = total oral intake in single consistency; 5 = total oral intake of multiple consistencies requiring special preparation; 6 = total oral intake with no special preparation, but must avoid specific foods or liquid items; 7 = total oral intake with no restrictions). A higher score is a better outcome.
Self-perceived swallowing impairment | Change in score from week 0 to week 5; change in score from week 0 to week 15; change in score from week 5 to week 15.
  Will be measured using the Eating Assessment Tool-10 (EAT-10), a self-administered, symptom-specific outcome instrument for dysphagia. The EAT-10 allows patients to rate their swallowing symptoms on scale of 0 = no problem to 4 = severe problem. A lower score is a better outcome.
Biomarker analyses | Baseline measurement (week 0)
  An optional blood sample will be collected for biomarker analysis, to identify correlations with clinical response. We will measure genetic biomarkers associated with swallowing function including rs6265, rs165599, rs10835211, rs17601696, and APOE4 genotype status. For these 5 genetic biomarkers, participants will be scored as having zero, one, or two alleles. This information will be used in subgroup analyses for the primary and secondary outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Pfeffer, MD, PhD, Principal Investigator — University of Calgary
Locations (1):
- Neuromuscular Clinic, South Health Campus, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ertekin C, Yuceyar N, Aydogdu, Karasoy H. Electrophysiological evaluation of oropharyngeal swallowing in myotonic dystrophy. J Neurol Neurosurg Psychiatry. 2001 Mar;70(3):363-71. doi: 10.1136/jnnp.70.3.363. PMID 11181860
- [Background] Luchesi KF, Kitamua S, Mourao LF. Amyotrophic Lateral Sclerosis survival analysis: Swallowing and non-oral feeding. NeuroRehabilitation. 2014;35(3):535-42. doi: 10.3233/NRE-141149. PMID 25238863
- [Background] Chio A, Logroscino G, Hardiman O, Swingler R, Mitchell D, Beghi E, Traynor BG; Eurals Consortium. Prognostic factors in ALS: A critical review. Amyotroph Lateral Scler. 2009 Oct-Dec;10(5-6):310-23. doi: 10.3109/17482960802566824. PMID 19922118
- [Background] Paris G, Martinaud O, Petit A, Cuvelier A, Hannequin D, Roppeneck P, Verin E. Oropharyngeal dysphagia in amyotrophic lateral sclerosis alters quality of life. J Oral Rehabil. 2013 Mar;40(3):199-204. doi: 10.1111/joor.12019. Epub 2012 Dec 27. PMID 23278936
- [Background] Yang R, Huang R, Chen D, Song W, Zeng Y, Zhao B, Zhou D, Shang HF. Causes and places of death of patients with amyotrophic lateral sclerosis in south-west China. Amyotroph Lateral Scler. 2011 May;12(3):206-9. doi: 10.3109/17482968.2011.572979. Epub 2011 Apr 21. PMID 21506897
- [Background] Abu-Baker A, Rouleau GA. Oculopharyngeal muscular dystrophy: recent advances in the understanding of the molecular pathogenic mechanisms and treatment strategies. Biochim Biophys Acta. 2007 Feb;1772(2):173-85. doi: 10.1016/j.bbadis.2006.10.003. Epub 2006 Oct 11. PMID 17110089
- [Background] Duranceau CA, Letendre J, Clermont RJ, Levesque HP, Barbeau A. Oropharyngeal dysphagia in patients with oculopharyngeal muscular dystrophy. Can J Surg. 1978 Jul;21(4):326-9. PMID 679079
- [Background] Pitts T, Bolser D, Rosenbek J, Troche M, Okun MS, Sapienza C. Impact of expiratory muscle strength training on voluntary cough and swallow function in Parkinson disease. Chest. 2009 May;135(5):1301-1308. doi: 10.1378/chest.08-1389. Epub 2008 Nov 24. PMID 19029430
- [Background] Troche MS, Okun MS, Rosenbek JC, Musson N, Fernandez HH, Rodriguez R, Romrell J, Pitts T, Wheeler-Hegland KM, Sapienza CM. Aspiration and swallowing in Parkinson disease and rehabilitation with EMST: a randomized trial. Neurology. 2010 Nov 23;75(21):1912-9. doi: 10.1212/WNL.0b013e3181fef115. PMID 21098406
- [Background] Silverman EP, Miller S, Zhang Y, Hoffman-Ruddy B, Yeager J, Daly JJ. Effects of expiratory muscle strength training on maximal respiratory pressure and swallow-related quality of life in individuals with multiple sclerosis. Mult Scler J Exp Transl Clin. 2017 May 29;3(2):2055217317710829. doi: 10.1177/2055217317710829. eCollection 2017 Apr-Jun. PMID 28607760
- [Background] Jones HN, Crisp KD, Robey RR, Case LE, Kravitz RM, Kishnani PS. Respiratory muscle training (RMT) in late-onset Pompe disease (LOPD): Effects of training and detraining. Mol Genet Metab. 2016 Feb;117(2):120-8. doi: 10.1016/j.ymgme.2015.09.003. Epub 2015 Sep 8. PMID 26381077
- [Background] Plowman EK, Tabor-Gray L, Rosado KM, Vasilopoulos T, Robison R, Chapin JL, Gaziano J, Vu T, Gooch C. Impact of expiratory strength training in amyotrophic lateral sclerosis: Results of a randomized, sham-controlled trial. Muscle Nerve. 2019 Jan;59(1):40-46. doi: 10.1002/mus.26292. Epub 2018 Nov 29. PMID 29981250
- [Background] Plowman EK, Watts SA, Tabor L, Robison R, Gaziano J, Domer AS, Richter J, Vu T, Gooch C. Impact of expiratory strength training in amyotrophic lateral sclerosis. Muscle Nerve. 2016 Jun;54(1):48-53. doi: 10.1002/mus.24990. Epub 2016 Mar 3. PMID 26599236
- [Background] Rosenbek JC, Robbins JA, Roecker EB, Coyle JL, Wood JL. A penetration-aspiration scale. Dysphagia. 1996 Spring;11(2):93-8. doi: 10.1007/BF00417897. PMID 8721066
- [Background] Nimmons D, Pendleton N, Payton A, Ollier W, Horan M, Wilkinson J, Hamdy S. A novel association between COMT and BDNF gene polymorphisms and likelihood of symptomatic dysphagia in older people. Neurogastroenterol Motil. 2015 Sep;27(9):1223-31. doi: 10.1111/nmo.12609. Epub 2015 Jun 14. PMID 26073434
- [Background] Raginis-Zborowska A, Pendleton N, Hamdy S. Genetic determinants of swallowing impairment, recovery and responsiveness to treatment. Curr Phys Med Rehabil Rep. 2016;4(4):249-256. doi: 10.1007/s40141-016-0133-6. Epub 2016 Aug 8. PMID 28018753
- [Background] Robison R, Tabor-Gray LC, Wymer JP, Plowman EK. Combined respiratory training in an individual with C9orf72 amyotrophic lateral sclerosis. Ann Clin Transl Neurol. 2018 Aug 21;5(9):1134-1138. doi: 10.1002/acn3.623. eCollection 2018 Sep. PMID 30250869
- [Background] Tabor LC, Rosado KM, Robison R, Hegland K, Humbert IA, Plowman EK. Respiratory training in an individual with amyotrophic lateral sclerosis. Ann Clin Transl Neurol. 2016 Sep 1;3(10):819-823. doi: 10.1002/acn3.342. eCollection 2016 Oct. PMID 27752517
- [Background] Belafsky PC, Mouadeb DA, Rees CJ, Pryor JC, Postma GN, Allen J, Leonard RJ. Validity and reliability of the Eating Assessment Tool (EAT-10). Ann Otol Rhinol Laryngol. 2008 Dec;117(12):919-24. doi: 10.1177/000348940811701210. PMID 19140539
- [Background] Crary MA, Mann GD, Groher ME. Initial psychometric assessment of a functional oral intake scale for dysphagia in stroke patients. Arch Phys Med Rehabil. 2005 Aug;86(8):1516-20. doi: 10.1016/j.apmr.2004.11.049. PMID 16084801
- [Background] Hutcheson KA, Barrow MP, Barringer DA, Knott JK, Lin HY, Weber RS, Fuller CD, Lai SY, Alvarez CP, Raut J, Lazarus CL, May A, Patterson J, Roe JW, Starmer HM, Lewin JS. Dynamic Imaging Grade of Swallowing Toxicity (DIGEST): Scale development and validation. Cancer. 2017 Jan 1;123(1):62-70. doi: 10.1002/cncr.30283. Epub 2016 Aug 26. PMID 27564246
- [Background] Plowman EK, Tabor LC, Robison R, Gaziano J, Dion C, Watts SA, Vu T, Gooch C. Discriminant ability of the Eating Assessment Tool-10 to detect aspiration in individuals with amyotrophic lateral sclerosis. Neurogastroenterol Motil. 2016 Jan;28(1):85-90. doi: 10.1111/nmo.12700. Epub 2015 Oct 28. PMID 26510823
- [Background] Chiara T, Martin AD, Davenport PW, Bolser DC. Expiratory muscle strength training in persons with multiple sclerosis having mild to moderate disability: effect on maximal expiratory pressure, pulmonary function, and maximal voluntary cough. Arch Phys Med Rehabil. 2006 Apr;87(4):468-73. doi: 10.1016/j.apmr.2005.12.035. PMID 16571384